CLINICAL TRIAL: NCT00640653
Title: HIV/Sexually Transmitted Disease (STD) Prevention Interventions for Black Adolescents
Brief Title: Efficacy of an Abstinence-Only HIV Risk-Reduction Intervention for Young African-American Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Jemmott, Kenneth B. Clark Professor of Communication and Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH062049 (NIH); R01MH062049 (NIH); DAHBR 9A-ASPA (Other: National Institute of Mental Health)
Record Dates: First submitted 2008-03-19; First posted 2008-03-21 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Sexual Behavior; Abstinence; Intervention Studies; HIV; Sexually Transmitted Infection; Theory of Planned Behavior; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Sexual Behavior | interventions — Natural Family Planning Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Abstinence-only (Experimental): Participants will receive the abstinence-only HIV/STD risk-reduction intervention.
  Interventions: Behavioral: Abstinence-only HIV/STD risk-reduction intervention
- Safer-sex only (Experimental): Participants will receive the safer-sex-only HIV/STD risk-reduction intervention.
  Interventions: Behavioral: Safer-sex-only HIV/STD risk-reduction intervention
- Comprehensive-long (Experimental): Participants will receive the 12-h long comprehensive HIV/STD risk-reduction intervention.
  Interventions: Behavioral: Long comprehensive HIV/STD risk-reduction intervention
- Comprehensive-short (Experimental): Participants will receive the 8-h short comprehensive HIV/STD risk-reduction intervention.
  Interventions: Behavioral: Short comprehensive HIV/STD risk-reduction intervention
- Health-promotion control (Active Comparator): Participants will receive the health promotion control intervention.
  Interventions: Behavioral: Health promotion control intervention

INTERVENTIONS:
Behavioral: Abstinence-only HIV/STD risk-reduction intervention — Participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence. The intervention is not an abstinence-until-marriage intervention; the target behavior is abstaining from sexual activity until later in life when the adolescent is more prepared to handle the consequences. The intervention does not contain inaccurate information, portray sex in a negative light, or employ a moralistic tone. It is not designed to affect condom use.
  Other Names: Abstinence
  Arms: Abstinence-only
Behavioral: Safer-sex-only HIV/STD risk-reduction intervention — Participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for using condoms during sexual intercourse. The intervention is not designed to influence abstinence.
  Other Names: Condom-use intervention
  Arms: Safer-sex only
Behavioral: Long comprehensive HIV/STD risk-reduction intervention — Participants will attend three sessions consisting of twelve 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence and for using condoms if participants decide to be sexually active. The intervention consists of the safer-sex-specific content (4 hours), the abstinence-specific content (4 hours), and the general content that is common to both of the single-component interventions (4 hours).
  Other Names: Abstinence and condom-use intervention; Abstinence-plus intervention
  Arms: Comprehensive-long
Behavioral: Short comprehensive HIV/STD risk-reduction intervention — Participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence and for using condoms if participants decide to be sexually active.
  Other Names: Abstinence and condom-use intervention; Abstinence-plus intervention
  Arms: Comprehensive-short
Behavioral: Health promotion control intervention — Participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for avoiding cigarette smoking and for incorporating a healthful diet, aerobic exercise, and breast and testicular self-examinations. The control intervention will focus on reducing risk of heart disease, hypertension, diabetes, and certain cancers. The intervention provides a control for "Hawthorne effects" to reduce the likelihood that the HIV/STD interventions' effects can be attributed to group interaction and special attention.
  Other Names: Chronic disease prevention intervention
  Arms: Health-promotion control

SUMMARY:
This study will develop and evaluate the effectiveness of culturally appropriate HIV/sexually transmitted disease risk-reduction interventions in reducing sexual risk behavior among young African-American adolescents.

DETAILED DESCRIPTION:
Adolescents risk the negative consequences of early sexual involvement, including not only HIV, but other sexually transmitted diseases (STDs) and unintended pregnancies. Compared with older adults, young people, especially African-American young people, are at higher risk of acquiring an STD. Specifically, people 15 to 24 years of age acquire nearly 50% of all new STDs in the United States, but this age group represents only 25% of the sexually active population. Adolescents are especially vulnerable to STD infections because of a lack of education about proper condom use and consequences of sexual risk behaviors. Previous research has suggested that behavioral interventions can reduce adolescents' sexual behaviors tied to risk of acquiring STDs. Nevertheless, there is continuous debate over the appropriateness and effectiveness of different types of adolescent sexual-risk-reduction interventions, including abstinence education or comprehensive sexual education. Few studies have tested the long-term effectiveness of abstinence education, which emphasizes delaying sexual initiation for sexually inexperienced adolescents. This study will compare the effectiveness of an abstinence-only HIV/STD risk-reduction intervention with other types of interventions in reducing sexual risk behavior among young African-American adolescents.

Participation in this study will last 24 months. Participants at participating schools will be randomly assigned to one of five treatment groups:

* Abstinence-only group participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence. This is not an abstinence-until-marriage intervention; the target behavior is abstaining from sexual activity until later in life when the adolescent is more prepared to handle the consequences. The intervention is not designed to affect condom use.
* Safer-sex-only group participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for using condoms during sexual intercourse. The intervention is not designed to influence abstinence.
* Long comprehensive group participants will attend three sessions consisting of twelve 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence and for using condoms if participants decide to be sexually active. The intervention will consist of 4 hours each of the safer-sex-specific content, the abstinence-specific content, and the general content that is common to both of the single-component interventions.
* Short comprehensive group participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence and for using condoms if participants decide to be sexually active.
* Health promotion control participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for avoiding cigarette smoking and for incorporating a healthful diet, aerobic exercise, and breast and testicular self-examinations. The control intervention will focus on reducing risk of heart disease, hypertension, diabetes, and certain cancers.

Sessions for all groups will be led by trained adult facilitators and will include group discussions, videos, games, brainstorming, experiential exercises, and skill-building activities designed to be educational, interactive, and entertaining. All participants will complete self-reports concerning sexual behaviors, condom use, and knowledge about STDs at baseline and Months 3, 6, 12, 18, and 24 of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Grade 6 or 7 student at a participating school
* Written parent or guardian consent to participate
* Self-identifies as African American or black

Exclusion Criteria:

- Those not meeting inclusion criteria were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2001-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B. Jemmott III, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Jemmott JB 3rd, Jemmott LS, Fong GT. Efficacy of a theory-based abstinence-only intervention over 24 months: a randomized controlled trial with young adolescents. Arch Pediatr Adolesc Med. 2010 Feb;164(2):152-9. doi: 10.1001/archpediatrics.2009.267. PMID 20124144
- [Result] Zhang J, Jemmott JB 3rd, Jemmott LS. Mediation and moderation of an efficacious theory-based abstinence-only intervention for African American adolescents. Health Psychol. 2015 Dec;34(12):1175-84. doi: 10.1037/hea0000244. Epub 2015 Jul 27. PMID 26214076

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive-long: Participants will receive the long comprehensive HIV/STD risk-reduction intervention.
  Long comprehensive HIV/STD risk-reduction intervention: Participants will attend three sessions consisting of twelve 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence and for using condoms if participants decide to be sexually active. The intervention consists of the safer-sex-specific content (4 hours), the abstinence-specific content (4 hours), and the general content that is common to both of the single-component interventions (4 hours).
- Comprehensive-short: Participants will receive the short comprehensive HIV/STD risk-reduction intervention.
  Short comprehensive HIV/STD risk-reduction intervention: Participants will attend two sessions consisting of eight 1-hour modules that are designed to increase knowledge, motivation, and skill for practicing abstinence and for using condoms if participants decide to be sexually active.
Period: Overall Study
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Started | 131 | 134 | 129 | 134 | 134
Followed-up at 3 mo | 126 | 127 | 125 | 129 | 126
Followed-up at 6 mo | 127 | 130 | 124 | 130 | 125
Followed-up at 12 mo | 124 | 121 | 115 | 122 | 116
Followed-up at 18 mo | 118 | 112 | 113 | 117 | 117
Followed-up at 24 mo | 114 | 116 | 105 | 112 | 112
Completed | 128 | 131 | 129 | 132 | 129
Not Completed | 3 | 3 | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Sociodemographic Characteristics and Self-Reported Sexual Behaviors at Baseline of Participating African American Students in Grades 6 and 7 by Intervention Arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control | Total
Number analyzed (Participants) | 131 | 134 | 129 | 134 | 134 | 662
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (0.8) | 11.9 (0.8) | 11.9 (0.8) | 12.0 (0.8) | 12.0 (0.8) | 12.0 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 70 | 70 | 73 | 354
  Male | 62 | 62 | 59 | 64 | 61 | 308
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 131 | 134 | 129 | 134 | 134 | 662
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 131 | 134 | 129 | 134 | 134 | 662
Grade in School [Number; unit: participants]
  7th | 68 | 71 | 73 | 77 | 77 | 366
  8th | 63 | 63 | 56 | 57 | 57 | 296
Live with both parents [Number; unit: participants]
  Yes | 46 | 46 | 40 | 43 | 46 | 221
  No | 85 | 88 | 89 | 91 | 88 | 441
Ever had sexual intercourse [Number; unit: participants]
  Yes | 31 | 28 | 32 | 27 | 35 | 153
  No | 100 | 106 | 97 | 107 | 99 | 509

OUTCOME MEASURES:

1. Primary Outcome: Self-report of Ever Having Sexual Intercourse
Description: Self-reported sexual initiation during the follow-up period among participants who reported never having sexual intercourse at baseline.
Time Frame: 24 months post-intervention
Population: Participants reporting never having sexual intercourse at baseline (i.e., virgins) with follow-up data on self-reported sexual intercourse during the post-intervention assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Number analyzed (Participants) | 92 | 97 | 85 | 95 | 88
Participants | 39 | 40 | 44 | 31 | 41
Statistical Analysis 1: Comparison: Abstinence-only vs Health-promotion Control; With alpha = .05, 2-tailed, and 37.4% of the control group initiating sexual intercourse by 24-month follow-up, a total sample size of 563 participants completing the trial was projected to provide power of 80% to detect a difference of 16.8% in self-reported sexual intercourse between an HIV intervention condition and the health promotion control condition; Test type: Superiority or Other; p = .03, generalized linear regression — The significance criterion was set at alpha = .05; Log link was specified; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.48 to 0.96] — Treatment was coded as 1 vs health control coded as 0

2. Secondary Outcome: Self-reported Sexual Intercourse in the Past 3 Months
Description: Self-report of having sexual intercourse in the past 3 months
Time Frame: Measured at baseline and 3, 6, 12, 18, and 24 months post-intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Number analyzed (Participants) | 127 | 130 | 128 | 131 | 129
Participants
  Baseline | 14 | 13 | 15 | 16 | 18
  3 months: number analyzed (Participants) | 125 | 126 | 124 | 129 | 126
  3 months | 12 | 19 | 22 | 15 | 26
  6 months: number analyzed (Participants) | 127 | 130 | 122 | 130 | 125
  6 months | 18 | 19 | 21 | 13 | 27
  12 months: number analyzed (Participants) | 124 | 121 | 115 | 121 | 116
  12 months | 24 | 33 | 34 | 27 | 25
  18 months: number analyzed (Participants) | 118 | 112 | 113 | 117 | 117
  18 months | 32 | 32 | 40 | 39 | 35
  24 months: number analyzed (Participants) | 114 | 116 | 105 | 112 | 112
  24 months | 35 | 38 | 42 | 33 | 42

3. Secondary Outcome: Self-report of Having Multiple Sexual Partners in the Past 3 Months
Description: Self-report of having sexual intercourse with more than one partner in the pat 3 months.
Time Frame: Measured at baseline and 3, 6, 12, 18, and 24 months post-intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Number analyzed (Participants) | 127 | 130 | 127 | 131 | 128
Participants
  Baseline | 11 | 9 | 6 | 4 | 10
  3 months: number analyzed (Participants) | 125 | 125 | 123 | 128 | 125
  3 months | 7 | 6 | 12 | 5 | 14
  6 months: number analyzed (Participants) | 126 | 128 | 121 | 129 | 124
  6 months | 7 | 6 | 7 | 4 | 18
  12 months: number analyzed (Participants) | 123 | 120 | 112 | 121 | 114
  12 months | 13 | 9 | 14 | 11 | 10
  18 months: number analyzed (Participants) | 117 | 111 | 110 | 114 | 116
  18 months | 9 | 16 | 17 | 21 | 17
  24 months: number analyzed (Participants) | 114 | 115 | 100 | 111 | 111
  24 months | 16 | 13 | 17 | 14 | 17

4. Secondary Outcome: Self-reported Consistent Condom Use in the Past 3 Months
Description: Self-report of using a condom during every sexual intercourse act in the past 3 months
Time Frame: Measured at baseline and 3, 6, 12, 18, and 24 months post-intervention
Population: Participants with data at baseline and at least one post intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Number analyzed (Participants) | 53 | 54 | 63 | 52 | 59
Participants
  Baseline: number analyzed (Participants) | 10 | 12 | 14 | 11 | 17
  Baseline | 7 | 8 | 4 | 10 | 12
  3-Months: number analyzed (Participants) | 13 | 18 | 21 | 15 | 25
  3-Months | 8 | 15 | 16 | 12 | 20
  6-Months: number analyzed (Participants) | 17 | 18 | 20 | 13 | 26
  6-Months | 14 | 17 | 17 | 11 | 15
  12-Months: number analyzed (Participants) | 23 | 31 | 34 | 26 | 24
  12-Months | 16 | 25 | 24 | 19 | 17
  18-Months: number analyzed (Participants) | 30 | 32 | 40 | 39 | 34
  18-Months | 23 | 21 | 34 | 31 | 27
  24-Months: number analyzed (Participants) | 35 | 37 | 42 | 33 | 41
  24-Months | 26 | 29 | 31 | 25 | 32

5. Secondary Outcome: Self-report of Having Sexual Intercourse Without Using a Condom During the Past 3 Months
Time Frame: Measured at baseline and3, 6, 12, 18, and 24 months post-intervention
Population: Participants with data at baseline and at least one post intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Number analyzed (Participants) | 127 | 129 | 127 | 131 | 129
Participants
  Baseline | 3 | 2 | 7 | 1 | 5
  3-Months: number analyzed (Participants) | 125 | 124 | 123 | 127 | 126
  3-Months | 5 | 2 | 4 | 1 | 4
  6-Months: number analyzed (Participants) | 125 | 128 | 122 | 128 | 125
  6-Months | 2 | 1 | 3 | 1 | 11
  12-Months: number analyzed (Participants) | 123 | 119 | 109 | 121 | 116
  12-Months | 7 | 6 | 6 | 7 | 7
  18-Months: number analyzed (Participants) | 117 | 109 | 108 | 116 | 117
  18-Months | 6 | 10 | 3 | 8 | 7
  24-Months: number analyzed (Participants) | 113 | 113 | 101 | 111 | 110
  24-Months | 8 | 8 | 8 | 8 | 8

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Comprehensive-long | Comprehensive-short | Safer-sex Only | Abstinence-only | Health-promotion Control
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/134 | 0/129 | 0/134 | 0/134
Other Adverse Events (participants affected / at risk) | 0/131 | 0/134 | 0/129 | 0/134 | 0/134

LIMITATIONS AND CAVEATS:
The data were based on self-reports, which can be inaccurate because of poor memory or socially desirability bias. The results may be limited to African American grade 6 and 7 students willing to take part in a health program on weekends.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No